CLINICAL TRIAL: NCT05447598
Title: Individually Tailored Remote Monitoring at Home After Hospitalisation for HEART Failure in Multi-morbid Patients (IT-HEART): a Randomised Clinical Trial
Brief Title: Remote Monitoring After Heart Failure
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vestre Viken Hospital Trust (Other)
Collaborators: The Hospital of Vestfold (Other); University of Oslo (Other); Oslo University Hospital (Other); University of Stavanger (Other); University Hospital, Akershus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 464460
Record Dates: First submitted 2022-05-27; First posted 2022-07-07 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure Acute; Remote Monitoring; Nurse's Role

STUDY DESIGN:
Intervention Model Description: Participants were randomized 1:1 to a nurse-led remote monitoring program or to usual care
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Remote monitoring program
  Interventions: Other: Nurse-led remote monitoring program
- Usual care (Active Comparator): Current clinical pratice at the participating hospitals
  Interventions: Other: Usual care treatment

INTERVENTIONS:
Other: Nurse-led remote monitoring program — Symptoms of disease progression, clinical parameters, medication adherence and follow-up needs will be reported by patients or with support from relatives or homecare nurses 2-4 times/months over a three months period using a digital platform. Telephone monitoring is planned for patients who are not able to comply with the digital platform. In addition, an individualized self-treatment plan for diuretics and lifestyle advice will be prepared, preferably together with relatives at the outpatient clinic. Participants will also have access to a website with written information and videos about HF and self-management. Finally, a pillbox will be delivered to facilitate drug adherence.
  Arms: Intervention
Other: Usual care treatment — Usual care treatment and follow-up care at the outpatient clinic and in primary care
  Arms: Usual care

SUMMARY:
Heart failure (HF) is a leading cause of hospitalisation and disability-adjusted life years lost, with mortality rates exceeding most cancers. Despite compelling evidence and recommendations, less than 20% of the HF patients are followed-up by the specialist healthcare after hospital discharge. Due to limited outpatient capacity, human resources and increasing incidence of HF over the next decades, new care models are obviously needed. Remote monitoring (i.e. telemonitoring) encompasses the use of audio, video and other telecommunication technologies to monitor patient status at a distance. Remote monitoring is a promising strategy that can facilitate rapid access to care when needed and reduce patient travel to hospital consultations. It also promotes self-care behaviour, psychosocial support, and early detection of cardiac decompensation. Despite intensive research for >10 years, randomised trials show conflicting results, and European HF guidelines are confined to a weak (class IIb, level of evidence B) recommendation. More knowledge about the role of remote monitoring strategies in HF management, especially in the transition from hospital to home, is thus requested in the most recent European and US guidelines. In particular, studies of high-risk patients integrating the community health services are largely lacking. Furthermore, the components of the intervention that mediate the effect need to be identified. The proposed study aims to address these gaps in evidence and assess whether individually tailored remote monitoring at home (IT-HEART) is improves clinical outcomes in patients hospitalized with decompensated HF. We also aim to identify modifiable clinical and behavioural (drug adherence, self-care, psychological factors) outcome predictors. A prospective, multicentre, randomized, open-label, blinded endpoint adjudication (PROBE) intervention study is designed and powered to include at least 200 patients with at least one HF hospitalization in the 12 months preceding enrolment. To ensure generalizability, patients will be included regardless of comorbidity, frailty and ejection fraction. We have conducted a pilot-study providing empirical evidence for the expected participation rate, readmission rate and barriers to HF management in current clinical practice that will be targets for the intervention. This will promote high adherence to the intervention and positive long-term clinical and health economic effects.

ELIGIBILITY:
Inclusion Criteria:

* Age> 18 years
* Known HF diagnosis (ICD-10: I50) recorded in hospital medical records
* Admitted to hospital within 7 days before screening for acute HF with symptoms of decompensation including dyspnoea in NYHA class ≥ II, pulmonary congestion on chest x-ray and/or other signs like oedema or positive rales on auscultation and elevated NT-proBNP concentrations at screening
* Sign informed consent and expected to participate according to ICH / GCP

Exclusion Criteria:

* Any condition (e.g. psychosis, alcohol abuse, dementia) or situation that may pose a significant risk to the participant, confuse the results or make participation unethical
* Not able to understand Norwegian language
* Short life expectancy (<6 months) due to non-cardiac causes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of re-hospitalizations for heart failure | From time of randomization until 12 months follow-up
  Rate of re-hospitalizations for heart failure at 12 months follow-up assessed from hospital medical records between the treatment arms
Time to first re-hospitalization for heart failure | From time of randomization until 12 months follow-up
  Time to first re-hospitalization for heart failure at 12 months follow-up assessed from hospital medical records between the treatment arms

SECONDARY OUTCOMES:
Rate of total death | From time of randomization until 12 months follow-up
  Rate of total death at 12 months follow-up assessed from hospital medical records between the treatment arms
Rate of unplanned re-hospitalizations | From time of randomization until 12 months follow-up
  Rate of re-hospitalizations at 12 months follow-up assessed from hospital medical records between the treatment arms
Total number of days lost due to unplanned heart failure admissions treatment arms | From time of randomization until 12 months follow-up
  Percentage of days lost due to unplanned heart failure admissions at 12 months follow-up between the treatment arms assessed from hospital medical records
Total number of days lost due to unplanned hospital admissions treatment arms | From time of randomization until 12 months follow-up
  Percentage of days lost due to unplanned hospital admissions at 12 months follow-up between the treatment arms assessed from hospital medical records
Changes in selfcare behaviour | From baseline until three months follow-up
  Changes in selfcare behaviour measured by the revised 9-item European Heart Failure Selfcare behaviour Scale assessed by patient self-report on a five-point scale from "totally agree" to "totally disagree".
Changes in health-related quality of life | From baseline until three months follow-up
  Changes in health-related quality of life measured by Kansas Cardiomyopathy Questionnaire 12-score (higher scores indicating better outcome).
Changes in symptom score and patient satisfaction | From baseline until three months follow-up
  Changes in symptom score and patient satisfaction measured by the Edmonton Symptom Assessment System Revised scores (higher scores indicating better outcome).

CONTACTS AND LOCATIONS:
Locations (3):
- Norway (3):
  - Vestfold Hospital Trust, Tønsberg, Vestfold and Telemark County
  - Vestre Viken Trust Drammen hospital, Drammen, Viken County
  - Akershus University Hospital, Lørenskog